CLINICAL TRIAL: NCT06157385
Title: The Effect of Culinary Medicine to Enhance Protein Intake on Muscle Quality in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB2023-505
Record Dates: First submitted 2023-10-26; First posted 2023-12-05 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia
Keywords: Culinary medicine; Protein intake; Muscle quality; Older adults
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culinary Medicine (Experimental): The participants in this group will receive culinary medicine in the form of videos that will include cooking demonstrations and nutrition education based on lean beef to enhance protein intake.
  Interventions: Behavioral: Culinary Medicine
- Control (Other): This group will only receive recipes based on lean beef to enhance protein intake.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Culinary Medicine — The CM group will receive virtually-delivered cooking demonstration videos every week and nutrition education videos every other week. The cooking demonstrations will provide them with visual instructions on how to incorporate lean beef into their diet. The nutrition education videos will be developed using the Nutrition Care Manual from the Academy of Nutrition and Dietetics and will cover the importance of maintaining adequate protein intake and ways to enhance it in the diet.
  Other Names: CM
  Arms: Culinary Medicine
Behavioral: Control — The CN group will receive virtually-delivered recipes every week centered on lean beef intake.
  Other Names: CN
  Arms: Control

SUMMARY:
Aging is associated with a decline in muscle mass, strength, and physical function, leading to sarcopenia and frailty. This deterioration of muscle and physical capabilities impacts an individual's functional independence and quality of life. Dietary protein stimulates muscle protein synthesis. Therefore, nutritional interventions that recommend higher protein intakes may enhance muscle protein synthesis. Food intake, including protein-rich foods such as red meat, has been shown to decline with age. Barriers to consuming protein-rich foods include reductions in taste and smell, dentition and dexterity, and changes in living situations. Therefore, nutritional interventions that can effectively improve eating behaviors and diet quality while stimulating muscle protein synthesis in older adults are necessary to help prevent, manage, and promote recovery of sarcopenia. To reduce potential barriers of red meat consumption in community-dwelling older adults, an additional beneficial strategy may be the use of cooking demonstrations, or culinary medicine, by imparting knowledge about healthy cooking to improve the dietary habits of individuals who are at risk of sarcopenia. In this approach, people will be educated about age-appropriate, healthy eating behaviors and equipped with basic cooking skills to incorporate nutritious food into their daily diet. A systematic review concluded that culinary interventions such as cooking classes effectively improved attitudes, self-efficacy, and healthy eating in children and adults. A recent study using cooking videos to encourage the consumption of calcium-rich foods showed that the subjects gained knowledge and were motivated to consume calcium-rich foods, and video demonstrations were accepted as an effective communication channel to impart cooking skills. Additionally, it is suggested that cooking at home improves adherence to healthy nutrition, thereby reducing chronic illness risks. Older adults may not be aware of their changing nutrient needs and therefore may lack the skills to prepare nutritionally adequate foods properly. Thus, cooking demonstrations can be a novel strategy to improve diet quality in older adults and promote and augment at-home cooking. Culinary medicine is an evidence-based field that combines skills of preparing, cooking, and presenting food with the science of medicine to accomplish potential improvements in eating behaviors and health outcomes. The goal of culinary medicine is to help people improve their diet quality which assists them in their medical regimen to produce an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* Physically active
* Willing to eat beef
* Able to cook
* Able to use a computer or mobile device
* Willing to undergo two blood draws

Exclusion Criteria:

* <65 years of age
* Screening for sarcopenia SARC-F score of 4 or greater
* Regular consumption of nicotine, excessive alcohol (4+ drinks/day for women or 5+ drinks/day for men), and/or illicit drugs such as amphetamines, cocaine, marijuana, or opiates
* Have cancer, transplant, amputation, or renal disorder
* Limited mobility
* Self-reported cognitive dysfunction
* Have heart pacemaker
* Have Type 1 diabetes or Type 2 diabetes with insulin therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Food Frequency Questionnaire (FFQ) | This will be assessed at baseline and after the 4-month intervention.
  The Diet History Questionnaire III (DHQ III) is a comprehensive FFQ that will be used to measure the subjects' protein intake and healthy eating index (HEI) for diet quality. The HEI uses a scoring system to evaluate a set of foods. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations and dietary patterns published in the Dietary Guidelines.
Weekly Cooking Effectiveness and Protein Intake Questionnaire | This will be assessed every week throughout the 4-month intervention starting at the end of the first week.
  This is a brief weekly questionnaire designed by the research team to assess the subjects' protein intake as well as their experience with the beef and culinary medicine or recipes that received for that week. There is no scale associated with this measurement. The researchers will evaluate the answers individually.

SECONDARY OUTCOMES:
Cooking Effectiveness Questionnaire | This will be assessed at baseline and after the 4-month intervention.
  This detailed questionnaire designed by the research team will assess the subjects' confidence, attitudes, and any possible barriers around cooking for themselves. There is no scale associated with this measurement. The researchers will evaluate the answers individually.
Nutrition Knowledge Questionnaire | This will be assessed at baseline and after the 4-month intervention.
  This questionnaire designed by the research team will assess the subjects' understanding of the nutritional qualities of red meat and other protein sources. This information will be used to gauge the effectiveness of the nutrition education provided. There is no scale associated with this measurement. The researchers will evaluate the answers individually.
Physical Activity Questionnaire | This will be assessed at baseline and after the 4-month intervention.
  The Physical Activity Scale for the Elderly (PASE) is a validated questionnaire for older adults that will be used to assess the physical activity rates of the subjects. There is no scale associated with this measurement. The researchers will evaluate the answers individually.
Handgrip Strength | This will be assessed at baseline and after the 4-month intervention.
  A handgrip dynamometer will be used to assess the muscle strength of the subjects. Their grip strengths will be measured three times with each hand, so an average of those three measurements can be calculated.
Short Physical Performance Battery (SPPB) Exam | This will be assessed at baseline and after the 4-month intervention.
  This is a validated test proctored by a member of the research team that consists of a series of exercises to assess the muscle function of the subjects. The scale is a minimum of 0 and maximum of 12 points overall.
Serum Value of Vitamin B12 in pg/mL | This will be assessed at baseline and after the 4-month intervention.
  A blood draw will be completed by a professional phlebotomist, and the sample collected will be analyzed to measure serum levels of vitamin B12. This nutrient is used in the process of muscle protein synthesis in the body and will be indicator of this process in the subjects.
Serum Value of Folate in ng/mL | This will be assessed at baseline and after the 4-month intervention.
  A blood draw will be completed by a professional phlebotomist, and the sample collected will be analyzed to measure serum levels of folate. This nutrient is used in the process of muscle protein synthesis in the body and will be indicator of this process in the subjects.
Serum Value of Creatinine in mg/dL | This will be assessed at baseline and after the 4-month intervention.
  A blood draw will be completed by a professional phlebotomist, and the sample collected will be analyzed to measure serum levels of creatinine. This nutrient is used in the process of muscle protein synthesis in the body and will be indicator of this process in the subjects.
Daily Steps | This will be collected throughout the study and assessed after the intervention.
  The subjects will be given a physical activity watch, the Garmin Vivofit 4, and instructed to wear it throughout each day for the duration of the study. This watch will collect the daily steps throughout the study and will be used to further assess physical activity rates of the subjects.
BMI in (lb/in^2)*703 | This will be assessed at baseline and after the 4-month intervention.
  This will be calculated with the Tanita MC-780U BIA Scale.
Weight in Pounds | This will be assessed at baseline and after the 4-month intervention.
  This will be measured using the Tanita MC-780U BIA Scale.
Height in Inches | This will be assessed at baseline and after the 4-month intervention.
  This will be measured using a stadiometer.
Muscle Composition with Bioelectric Impedance Analysis (BIA) Tanita MC-780U Scale | This will be assessed at baseline and after the 4-month intervention.
  This will assess the muscle mass which will give an indication of muscle composition.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Galyean, Principal Investigator — Texas Tech Nutritional Sciences
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Porter Starr KN, Orenduff M, McDonald SR, Mulder H, Sloane R, Pieper CF, Bales CW. Influence of Weight Reduction and Enhanced Protein Intake on Biomarkers of Inflammation in Older Adults with Obesity. J Nutr Gerontol Geriatr. 2019 Jan-Mar;38(1):33-49. doi: 10.1080/21551197.2018.1564200. Epub 2019 Feb 27. PMID 30810500
- [Background] Hengeveld LM, Boer JMA, Gaudreau P, Heymans MW, Jagger C, Mendonca N, Ocke MC, Presse N, Sette S, Simonsick EM, Tapanainen H, Turrini A, Virtanen SM, Wijnhoven HAH, Visser M. Prevalence of protein intake below recommended in community-dwelling older adults: a meta-analysis across cohorts from the PROMISS consortium. J Cachexia Sarcopenia Muscle. 2020 Oct;11(5):1212-1222. doi: 10.1002/jcsm.12580. Epub 2020 Jun 16. PMID 32548960
- [Background] Viitasalo JT, Era P, Leskinen AL, Heikkinen E. Muscular strength profiles and anthropometry in random samples of men aged 31-35, 51-55 and 71-75 years. Ergonomics. 1985;28(11):1563-74.
- [Background] Avlund K, Schroll M, Davidsen M, Løvborg B, Rantanen T. Maximal isometric muscle strength and functional ability in daily activities among 75-year-old men and women. Scandinavian Journal of Medicine & Science in Sports. 1994;4(1):32-40.
- [Background] Genaro Pde S, Martini LA. Effect of protein intake on bone and muscle mass in the elderly. Nutr Rev. 2010 Oct;68(10):616-23. doi: 10.1111/j.1753-4887.2010.00321.x. PMID 20883419
- [Background] Franzke B, Neubauer O, Cameron-Smith D, Wagner KH. Dietary Protein, Muscle and Physical Function in the Very Old. Nutrients. 2018 Jul 20;10(7):935. doi: 10.3390/nu10070935. PMID 30037048
- [Background] Ni Lochlainn M, Bowyer RCE, Steves CJ. Dietary Protein and Muscle in Aging People: The Potential Role of the Gut Microbiome. Nutrients. 2018 Jul 20;10(7):929. doi: 10.3390/nu10070929. PMID 30036990
- [Background] Cholewa JM, Dardevet D, Lima-Soares F, de Araujo Pessoa K, Oliveira PH, Dos Santos Pinho JR, Nicastro H, Xia Z, Cabido CE, Zanchi NE. Dietary proteins and amino acids in the control of the muscle mass during immobilization and aging: role of the MPS response. Amino Acids. 2017 May;49(5):811-820. doi: 10.1007/s00726-017-2390-9. Epub 2017 Feb 7. PMID 28175999
- [Background] Jyvakorpi SK, Pitkala KH, Puranen TM, Bjorkman MP, Kautiainen H, Strandberg TE, Soini H, Suominen MH. Low protein and micronutrient intakes in heterogeneous older population samples. Arch Gerontol Geriatr. 2015 Nov-Dec;61(3):464-71. doi: 10.1016/j.archger.2015.06.022. Epub 2015 Jul 15. PMID 26298429
- [Background] Berner LA, Becker G, Wise M, Doi J. Characterization of dietary protein among older adults in the United States: amount, animal sources, and meal patterns. J Acad Nutr Diet. 2013 Jun;113(6):809-15. doi: 10.1016/j.jand.2013.01.014. Epub 2013 Mar 13. PMID 23491327
- [Background] Fulgoni VL 3rd. Current protein intake in America: analysis of the National Health and Nutrition Examination Survey, 2003-2004. Am J Clin Nutr. 2008 May;87(5):1554S-1557S. doi: 10.1093/ajcn/87.5.1554S. PMID 18469286
- [Background] Appleton KM. Barriers to and Facilitators of the Consumption of Animal-Based Protein-Rich Foods in Older Adults. Nutrients. 2016 Mar 29;8(4):187. doi: 10.3390/nu8040187. PMID 27043615
- [Background] LeBlanc-Morales N. Culinary Medicine: Patient Education for Therapeutic Lifestyle Changes. Crit Care Nurs Clin North Am. 2019 Mar;31(1):109-123. doi: 10.1016/j.cnc.2018.11.009. Epub 2018 Dec 24. PMID 30736931
- [Background] La Puma J. What Is Culinary Medicine and What Does It Do? Popul Health Manag. 2016 Feb;19(1):1-3. doi: 10.1089/pop.2015.0003. Epub 2015 Jun 2. No abstract available. PMID 26035069
- [Background] Hasan B, Thompson WG, Almasri J, Wang Z, Lakis S, Prokop LJ, Hensrud DD, Frie KS, Wirtz MJ, Murad AL, Ewoldt JS, Murad MH. The effect of culinary interventions (cooking classes) on dietary intake and behavioral change: a systematic review and evidence map. BMC Nutr. 2019 May 10;5:29. doi: 10.1186/s40795-019-0293-8. eCollection 2019. PMID 32153942
- [Background] Bramston V, Rouf A, Allman-Farinelli M. The Development of Cooking Videos to Encourage Calcium Intake in Young Adults. Nutrients. 2020 Apr 27;12(5):1236. doi: 10.3390/nu12051236. PMID 32349354
- [Background] Polak R, Tirosh A, Livingston B, Pober D, Eubanks JE Jr, Silver JK, Minezaki K, Loten R, Phillips EM. Preventing Type 2 Diabetes with Home Cooking: Current Evidence and Future Potential. Curr Diab Rep. 2018 Sep 14;18(10):99. doi: 10.1007/s11892-018-1061-x. PMID 30218282
- [Background] Wolfson JA, Leung CW, Richardson CR. More frequent cooking at home is associated with higher Healthy Eating Index-2015 score. Public Health Nutr. 2020 Sep;23(13):2384-2394. doi: 10.1017/S1368980019003549. Epub 2020 Jan 10. PMID 31918785
- [Background] Irl B H, Evert A, Fleming A, Gaudiani LM, Guggenmos KJ, Kaufer DI, McGill JB, Verderese CA, Martinez J. Culinary Medicine: Advancing a Framework for Healthier Eating to Improve Chronic Disease Management and Prevention. Clin Ther. 2019 Oct;41(10):2184-2198. doi: 10.1016/j.clinthera.2019.08.009. Epub 2019 Sep 20. PMID 31543284
- [Background] Zivkovic AM, German JB. Metabolomics for assessment of nutritional status. Curr Opin Clin Nutr Metab Care. 2009 Sep;12(5):501-7. doi: 10.1097/MCO.0b013e32832f1916. PMID 19584717
- [Background] Santarpia L, Contaldo F, Pasanisi F. Dietary protein content for an optimal diet: a clinical view. J Cachexia Sarcopenia Muscle. 2017 Jun;8(3):345-348. doi: 10.1002/jcsm.12176. Epub 2017 Apr 25. PMID 28444858
- [Background] Micha R, Michas G, Mozaffarian D. Unprocessed red and processed meats and risk of coronary artery disease and type 2 diabetes--an updated review of the evidence. Curr Atheroscler Rep. 2012 Dec;14(6):515-24. doi: 10.1007/s11883-012-0282-8. PMID 23001745
- [Background] Micha R, Wallace SK, Mozaffarian D. Red and processed meat consumption and risk of incident coronary heart disease, stroke, and diabetes mellitus: a systematic review and meta-analysis. Circulation. 2010 Jun 1;121(21):2271-83. doi: 10.1161/CIRCULATIONAHA.109.924977. Epub 2010 May 17. PMID 20479151
- [Background] O'Connor LE, Paddon-Jones D, Wright AJ, Campbell WW. A Mediterranean-style eating pattern with lean, unprocessed red meat has cardiometabolic benefits for adults who are overweight or obese in a randomized, crossover, controlled feeding trial. Am J Clin Nutr. 2018 Jul 1;108(1):33-40. doi: 10.1093/ajcn/nqy075. PMID 29901710
- [Background] Gilmore LA, Walzem RL, Crouse SF, Smith DR, Adams TH, Vaidyanathan V, Cao X, Smith SB. Consumption of high-oleic acid ground beef increases HDL-cholesterol concentration but both high- and low-oleic acid ground beef decrease HDL particle diameter in normocholesterolemic men. J Nutr. 2011 Jun;141(6):1188-94. doi: 10.3945/jn.110.136085. Epub 2011 Apr 27. PMID 21525253